CLINICAL TRIAL: NCT05009628
Title: Is Routine Postoperative Oxygen Therapy Still Necessary in 2020?
Acronym: FreeO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019_0006
Record Dates: First submitted 2021-08-06; First posted 2021-08-17 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Oxygen Therapy

STUDY DESIGN:
Intervention Model Description: interventional study with 4 paralel arms ; randomization is realised according to a centralized and balanced 2x2 factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- automated oxygenation with a sitting patient position in the ICU (Experimental)
  Interventions: Procedure: automated oxygenation with a sitting patient position in the ICU
- controlled oxygenation with a lying patient position in the ICU (No Intervention)
- automated oxygenation with the patient lying down in the ICU (Experimental)
  Interventions: Procedure: Automated oxygenation with the patient lying down in the ICU
- control oxygenation with the patient in a sitting position in the ICU (Experimental)
  Interventions: Procedure: Oxygenation is controlled with the patient in a sitting position in the ICU.

INTERVENTIONS:
Procedure: automated oxygenation with a sitting patient position in the ICU — Oxygenation will be done with the Free O2 device via oxygen goggles or a face mask and with an O2 prescription to obtain a SpO2> 94%. The patient's position in the ICU will be a sitting position with the chest raised at an angle greater than 45°.
  Arms: automated oxygenation with a sitting patient position in the ICU
Procedure: Automated oxygenation with the patient lying down in the ICU — Oxygenation will be done with the Free O2 device via oxygen goggles or a face mask and with an O2 prescription to obtain a SpO2> 94%. The patient's position in the ICU will be a recumbent position with the head elevated to a maximum of 10
  Arms: automated oxygenation with the patient lying down in the ICU
Procedure: Oxygenation is controlled with the patient in a sitting position in the ICU. — ICU. Oxygenation will be done via the same interface in manual mode where the post-interventional monitoring room nurse modifies the flow to maintain oxygen saturation above 94%. The patient's position in the ICU will be a sitting position with the chest raised at an angle greater than 45°.
  Arms: control oxygenation with the patient in a sitting position in the ICU

SUMMARY:
The purpose of this study by automated control of oxygen supply in the immediate postoperative period is to show the possibility of immediate weaning in the postoperative period in case of remifentanil use and complete reversion of curarization.

DETAILED DESCRIPTION:
The main hypothesis of this study is that classical oxygen therapy at 3l/min is futile in the postoperative period of a so-called modern anaesthesia and that a total weaning within one hour after arrival in the ICU is possible whatever the postoperative position of the patient. The aim is therefore to include patients who have to undergo a scheduled surgery under anaesthetic sedation (analgesia with remifentanil) or general anaesthesia (combining remifentanil, propofol rocuronium) for ambulatory surgery. The trial is interventional, randomized, monocentric to demonstrate the absence of interest of prolonged postoperative oxygen therapy under specific intraoperative conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients managed by the Anesthesia Department of the Foch Hospital;
* Anesthetic sedation (analgesia with remifentanil) or general anesthesia (combining remifentanil, propofol and possibly rocuronium);
* Men or women over 18 and under 80 years of age;
* To benefit from a surgical intervention scheduled > 48 hours in relation to the procedure;
* Scheduled outpatient surgery;
* Have signed a consent form;
* Be affiliated to a health insurance plan.

Exclusion Criteria:

* Pregnant or nursing patients;
* Oxygen dependent preoperatively or at risk of oxygen dependence postoperatively;
* Lung resection surgery;
* Brain surgery (intracerebral neurosurgery); ENT surgery requiring a half-seated position after the operation;
* Being deprived of liberty or under guardianship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Oxygen withdrawal time | 1 day
  Time (min) to achieve zero O2 flow for at least 15 consecutive minutes

SECONDARY OUTCOMES:
Amount of O2 needed to reach the target saturation value (SpO2) | 1 day
  Number of liters of O2 needed postoperatively
Rate of patients weaned within the first hour | 1 day
  Zero O2 flow for at least 15 consecutive minutes
Signature time in the ICU | 1 day
  Minutes since admission
Maximum flow rate during the evaluation period | 1 day
  Maximum value of O2 flow in liter/min
The patient's comfort | 1 day
  Numerical scale between 0 and 10 to evaluate patient comfort
Complications during hospital stay | 30 days
  Length of hospital stay
Complications during stay in intensive care unit | 30 days
  Length of stay in intensive care unit
Mortality during stay in hospital | 30 days
  Hospital mortality
Complications after stay in hospital | 30 days
  Rehospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Foch, Suresnes, France